CLINICAL TRIAL: NCT01020474
Title: A 15 Week, Randomized, Double Blind, Parallel-group, Placebo-controlled, Flexible-dose, Safety And Efficacy Study Of Pregabalin In Adolescents (12-17 Years Old) With Fibromyalgia
Brief Title: Adolescent Fibromyalgia Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081180; 2010-019521-34 (EudraCT Number)
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Results first posted 2015-06-25 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-06

CONDITIONS: Fibromyalgia
Keywords: juvenile primary fibromyalgia syndrome; pediatric fibromyalgia; pregabalin; and Lyrica
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- drug-pregabalin (Experimental)
  Interventions: Drug: pregabalin (Lyrica)

INTERVENTIONS:
Drug: placebo — matching placebo capsules twice daily.
  Arms: Placebo
Drug: pregabalin (Lyrica) — 75-450mg/day pregabalin dose optimised at start of study
  Arms: drug-pregabalin

SUMMARY:
This study will compare pregabalin with placebo over a 15 week period in adolescents with fibromyalgia aged 12-17 years to evaluate the safety and efficacy of pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* 12-17 years of age

Exclusion Criteria:

* Patients with other pain conditions
* Previous treatment with pregabalin
* Patients taking excluded medication

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 107 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (30):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Apex Research Institute, Santa Ana, California
  - Eileen Messing, Psy D., Delray Beach, Florida
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Delray Research Associates, Delray Beach, Florida
  - Florida Medical Center and Research, Inc., Miami, Florida
  - Harmony Clinical Research, Incorporated, North Miami Beach, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Medical Research & Health Education Foundation, Inc., Columbus, Georgia
  - North Georgia Rheumatology, PC, Lawrenceville, Georgia
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University Pediatric Rheumatology of Kentucky, LLC, Louisville, Kentucky
  - University of Massachusetts Memorial Medical Center Department of Pediatrics, Worcester, Massachusetts
  - A&A Pain Institute of St. Louis, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Duke Medicine Plaza, Raleigh, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Akron Children's Hospital, Boardman, Ohio
  - Boardman Medical Pavilion, Boardman, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - St. Christopher's Hospital for Children / Section of Rheumatology, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Pediatric Rheumatology, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC University Children's Hospital, Charleston, South Carolina
  - Carolina Research Center, Myrtle Beach, South Carolina
  - Fatigue Consultation Clinic, Salt Lake City, Utah
- Bioregeneracni a rehabilitacni centrum, Říčany, Czechia
- India (4):
  - Krishna Institute of Medical Sciences Ltd, Secunderabad, Andhra Pradesh
  - Mallikatta Neuro Centre, Mangalore, Karnataka
  - Sushrut Hospital, Research Centre & Post Graduate Institute of Orthopaedics, Nagpur, Maharashtra
  - Department of Physical Medicine & Rehabilitation, Lucknow, Uttar Pradesh
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Arnold LM, Schikler KN, Bateman L, Khan T, Pauer L, Bhadra-Brown P, Clair A, Chew ML, Scavone J; Pregabalin Adolescent Fibromyalgia Study Group. Safety and efficacy of pregabalin in adolescents with fibromyalgia: a randomized, double-blind, placebo-controlled trial and a 6-month open-label extension study. Pediatr Rheumatol Online J. 2016 Jul 30;14(1):46. doi: 10.1186/s12969-016-0106-4. PMID 27475753
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081180&StudyName=Adolescent%20Fibromyalgia%20Study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 147 participants were screened, 107 participants were randomized to treatment. The 107 randomized participants were recruited in 4 countries at 23 study centers.
Pre-assignment Details: This study consisted of 4 phases, screening (1 Week), dose optimization (3 Weeks), fixed dose (12 Weeks) and follow-up (1 Week).
Groups:
- Pregabalin: Pregabalin was administered orally, BID (twice a day) for 15 weeks (3 week dose optimization phase and 12 week fixed-dose phase). Participants received 75 milligram per day (mg/day) to 450 mg/day. Dosing was started on Day 1. The dose was optimized over a 3-week period followed by an additional 12 weeks at the optimized dose.
- Placebo: Placebo was administered orally, BID for 15 weeks (3 week dose optimization phase and 12 week fixed-dose phase). Dosing was started on Day 1.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 54 | 53
Completed | 44 | 36
Not Completed | 10 | 17
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Other Reasons | 1 | 1
Not completed — Insufficient Clinical Response | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Pregabalin was administered orally, BID for 15 weeks (3 week dose optimization phase and 12 week fixed-dose phase). Participants received 75 mg/day to 450 mg/day. Dosing was started on Day 1. The dose was optimized over a 3-week period followed by an additional 12 weeks at the optimized dose.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.2) | 14.7 (1.2) | 14.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 92
  Male | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 15 in Mean Pain Diary Score
Description: The Primary Endpoint is based on the daily pain diary, and is defined as change from baseline to Week 15 in mean pain diary score. The daily pain diary consists of an 11-point numeric rating scale ranging from zero (no pain) to 10 (worst possible pain). The patients rate their pain during the past 24 hours by choosing the appropriate number between 0 ("no pain") and 10 ("worst possible pain").
Time Frame: Week 15
Population: The full analysis set (FAS) population consists of all randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 51
Units on a scale | -1.60 (0.32) | -0.94 (0.31)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.121, ANCOVA — Missing data for week 15 mean pain score are imputed based on distribution of baseline pain scores if participants discontinue due to adverse events/ abnormal laboratory test results or lack of efficacy; Based on LS Means using analysis of covariance (ANCOVA) model (including Treatment, Center, Baseline value as covariate); Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.51 to 0.18]

2. Secondary Outcome: Change From Baseline to Week 15 in Mean Sleep Quality Diary Score
Description: Change from Baseline to endpoint in mean sleep quality score from the daily sleep diary, defined as the mean of the last 7 diary entries prior to Visit 10 in the study while the participant is on study medication. The daily quality of sleep diary consists of an 11-point numeric rating scale with which the patient rates the quality of their sleep during the past 24 hours. Zero indicates "best possible sleep" and 10 indicates "worst possible sleep".
Time Frame: Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication. Last observation carried forward (LOCF) for participants with missing Week 15 mean pain score, i.e., the endpoint mean pain score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 50
Units on a scale | -1.13 (0.30) | -0.94 (0.31)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.655, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.00 to 0.63]

3. Secondary Outcome: Mean Change From Baseline to Weekly Mean Pain Score - Daily Pain Numeric Rating Scale (NRS)
Description: Mean pain score was calculated for each week during the double-blind treatment phase (Week 1 to Week 15). For each week, only days up to the last day on study medication were considered. A minimum of 4 pain diaries were required to calculate the mean pain score. The pain NRS consists of an 11 point NRS ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline to Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 51
Units on a scale
  Week 1 (N= 52, 49) | -0.48 (0.25) | -0.41 (0.26)
  Week 2 (N= 54, 47) | -1.11 (0.25) | -0.48 (0.26)
  Week 3 (N= 52, 44) | -1.27 (0.25) | -0.45 (0.26)
  Week 4 (N= 50, 46) | -1.45 (0.25) | -0.55 (0.26)
  Week 5 (N= 49, 44) | -1.27 (0.25) | -0.59 (0.26)
  Week 6 (N= 49, 44) | -1.47 (0.25) | -0.51 (0.27)
  Week 7 (N= 48, 42) | -1.67 (0.25) | -0.77 (0.27)
  Week 8 (N= 46, 44) | -1.65 (0.25) | -0.59 (0.27)
  Week 9 (N= 46, 42) | -1.61 (0.26) | -0.66 (0.27)
  Week 10 (N= 45, 40) | -1.82 (0.26) | -0.85 (0.27)
  Week 11 (N= 44, 38) | -1.93 (0.26) | -1.07 (0.28)
  Week 12 (N= 43, 34) | -1.75 (0.26) | -0.78 (0.28)
  Week 13 (N= 42, 33) | -1.75 (0.27) | -1.01 (0.29)
  Week 14 (N= 41, 34) | -2.01 (0.27) | -1.11 (0.29)
  Week 15 (N= 35, 33) | -1.90 (0.28) | -1.16 (0.30)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 1; Test type: Superiority or Other; p = 0.842, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.75 to 0.61]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 2; Test type: Superiority or Other; p = 0.070, Mixed Models Analysis; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.32 to 0.05]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 3; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.51 to -0.14]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 4; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.59 to -0.21]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 5; Test type: Superiority or Other; p = 0.056, Mixed Models Analysis; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.38 to 0.02]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 6; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.66 to -0.26]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 7; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-1.60 to -0.19]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 8; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-1.77 to -0.35]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 9; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Median Difference (Final Values) = -0.95, 95% CI 2-sided [-1.67 to -0.24]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 10; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.69 to -0.25]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 11; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.59 to -0.13]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 12; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.71 to -0.23]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 13; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.49 to 0.00]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 14; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.66 to -0.14]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 15; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.51 to 0.03]

4. Secondary Outcome: Mean Change From Baseline to Weekly Mean Sleep Quality Score (NRS)
Description: Mean sleep quality score was calculated for each week during the double-blind treatment phase (Week 1 to Week 15). A minimum of 4 sleep diaries are required to calculate the mean pain score. The daily quality of sleep diary consists of an 11-point numeric rating scale with which the patient rates the quality of their sleep during the past 24 hours. Zero indicates "best possible sleep" and 10 indicates "worst possible sleep".
Time Frame: Baseline to Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 51
Units on a scale
  Week 1 (N= 52, 49) | -0.52 (0.25) | -0.30 (0.26)
  Week 2 (N= 54, 47) | -0.84 (0.25) | -0.65 (0.26)
  Week 3 (N= 52, 44) | -0.89 (0.25) | -0.44 (0.26)
  Week 4 (N= 50, 46) | -1.03 (0.25) | -0.54 (0.26)
  Week 5 (N= 49, 44) | -0.99 (0.25) | -0.61 (0.27)
  Week 6 (N= 49, 44) | -1.18 (0.25) | -0.54 (0.27)
  Week 7 (N= 48, 42) | -1.30 (0.25) | -0.81 (0.27)
  Week 8 (N= 46, 44) | -1.43 (0.25) | -0.42 (0.27)
  Week 9 (N= 46, 42) | -1.38 (0.26) | -0.81 (0.27)
  Week 10 (N= 45, 40) | -1.43 (0.26) | -0.66 (0.27)
  Week 11 (N= 44, 38) | -1.39 (0.26) | -0.95 (0.28)
  Week 12 (N= 43, 34) | -1.38 (0.26) | -0.77 (0.28)
  Week 13 (N= 42, 33) | -1.34 (0.27) | -1.00 (0.29)
  Week 14 (N= 41, 34) | -1.36 (0.27) | -0.94 (0.29)
  Week 15 (N= 35, 33) | -1.25 (0.28) | -1.08 (0.30)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 1; Test type: Superiority or Other; p = 0.540, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.90 to 0.47]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 2; Test type: Superiority or Other; p = 0.593, Mixed Models Analysis; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.87 to 0.50]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 3; Test type: Superiority or Other; p = 0.206, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.13 to 0.25]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 4; Test type: Superiority or Other; p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.18 to 0.21]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 5; Test type: Superiority or Other; p = 0.280, Mixed Models Analysis; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-1.08 to 0.32]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 6; Test type: Superiority or Other; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.34 to 0.06]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 7; Test type: Superiority or Other; p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.21 to 0.21]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 8; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-1.73 to -0.30]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 9; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis; Median Difference (Final Values) = -0.57, 95% CI 2-sided [-1.29 to 0.15]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 10; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.49 to -0.05]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 11; Test type: Superiority or Other; p = 0.246, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-1.16 to 0.30]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 12; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.36 to 0.13]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 13; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.09 to 0.41]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 14; Test type: Superiority or Other; p = 0.285, Mixed Models Analysis; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.18 to 0.35]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; Statistical analysis of Week 15; Test type: Superiority or Other; p = 0.663, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.95 to 0.61]

5. Secondary Outcome: Change From Baseline to Week 15 in Mean Pain Numeric Rating Scale (1 Week Recall Period)
Description: The weekly pain numeric rating scale (Weekly Pain NRS) consists of an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate greater degree of impairment. Participants choose the number that best describes the pain during the last week.
Time Frame: Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication. Baseline observation carried forward (BOCF) for participants with missing Week 15 mean pain score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 53
Units on a scale | -1.64 (0.31) | -0.77 (0.30)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.037, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.68 to -0.05]

6. Secondary Outcome: Proportion of 30% Responders in Weekly Mean Pain Score (NRS) at Week 15
Description: At each visit, participants with at least 30% reduction from Baseline in mean pain score were defined as a 30% responder at the visit. The pain NRS consists of an 11 point NRS ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication. Modified baseline observation carried forward (mBOCF) for participants with missing Week 15 mean pain score.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 49
percentage of participants | 42.6 | 38.8
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 15; Test type: Superiority or Other; p = 0.694, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.53 to 2.58]

7. Secondary Outcome: Proportion of 50% Responder in Weekly Mean Pain Score (NRS) at Week 15
Description: At each visit, participants with at least 50% reduction from Baseline in mean pain score were defined as a 50% responder at the visit. The pain NRS consists of an 11 point NRS ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication. mBOCF for participants with missing Week 15 mean pain score.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 54 | 49
percentage of participants | 20.4 | 10.2
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 15; Test type: Superiority or Other; p = 0.162, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.72 to 7.02]

8. Secondary Outcome: Proportion of Patient Global Impression Change (PGIC) at Week 15
Description: Responder rates based on PGIC was derived and tabulated by treatment group. A responder was defined as a participant who reports much improved or very much improved. The PGIC is a patient-rated single item that measures patient's perception of change in their overall status since starting study medication on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 15
Population: The FAS population consists of all randomized participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 49 | 44
percentage of participants
  Very much improved | 16.3 | 2.3
  Much improved | 36.7 | 27.3
  Minimally improved | 22.4 | 27.3
  No change | 18.4 | 38.6
  Minimally worse | 6.1 | 2.3
  Much worse | 0 | 2.3
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis at Week 15; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel; P-value uses the row mean score statistic based on Cochran Mantel Haenszel (CMH) test with modified ridit transformation

ADVERSE EVENTS:
Time Frame: Adverse events were reported from signing the informed consent until a follow-up visit (Week 16).
Description: Participants are only counted once per treatment for each event.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/54 | 0/53
Other Adverse Events (participants affected / at risk) | 33/54 | 27/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=54) | Placebo (N=53)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=54) | Placebo (N=53)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 12 | 5
Vomiting (Gastrointestinal disorders) | 3 | 4
Fatigue (General disorders) | 8 | 4
Pyrexia (General disorders) | 4 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0
Weight increased (Investigations) | 9 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Balance disorder (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 16 | 7
Headache (Nervous system disorders) | 10 | 10
Migraine (Nervous system disorders) | 2 | 3
Somnolence (Nervous system disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.